CLINICAL TRIAL: NCT05130060
Title: Phase Ib Open-Label Study to Evaluate Safety, Tolerability, Immunogenicity and Efficacy of Multiple Subcutaneous Injections of PolyPEPI1018 Vaccine as an Add-on Immunotherapy to TAS-102 in Late-Stage Metastatic Colorectal Cancer Subjects
Brief Title: A Vaccine (PolyPEPI1018 Vaccine) and TAS-102 for the Treatment of Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC200404; NCI-2021-11619 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CA190836 (Other Grant/Funding Number: Department of Defense); 20-013410 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2021-11-10; First posted 2021-11-22 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Metastatic Colon Adenocarcinoma; Metastatic Colorectal Adenocarcinoma; Metastatic Colorectal Carcinoma; Metastatic Microsatellite Stable Colon Carcinoma; Metastatic Microsatellite Stable Colorectal Carcinoma; Metastatic Rectal Adenocarcinoma; Microsatellite Stable Rectal Carcinoma; Stage IV Colorectal Cancer AJCC v8; Stage IVA Colorectal Cancer AJCC v8; Stage IVB Colorectal Cancer AJCC v8; Stage IVC Colorectal Cancer AJCC v8
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms; Rectal Neoplasms | interventions — Trifluridine; trifluridine tipiracil drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (PolyPEPI1018, TAS-102) (Experimental): Patients receive PolyPEPI1018 SC at 4 injection sites on days 1 and 15 and trifluridine and tipiracil hydrochloride PO BID on days 1-5 and 8-15. Treatment repeats every 28 days for up to 7 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Colorectal Cancer Peptide Vaccine PolyPEPI1018; Drug: Trifluridine and Tipiracil Hydrochloride

INTERVENTIONS:
Biological: Colorectal Cancer Peptide Vaccine PolyPEPI1018 — Given SC
  Other Names: PolyPEPI 1018; PolyPEPI-1018; PolyPEPI1018; PolyPEPI1018 CRC Peptide Vaccine; PolyPEPI1018 CRC Vaccine
Drug: Trifluridine and Tipiracil Hydrochloride — Given PO
  Other Names: Lonsurf; TAS 102; TAS-102; Tipiracil Hydrochloride Mixture with Trifluridine; Trifluridine/Tipiracil; Trifluridine/Tipiracil Hydrochloride Combination Agent TAS-102

SUMMARY:
This phase Ib trial studies the safety and side effects of a vaccine (PolyPEPI1018 vaccine) in combination with TAS-102 in treating patients with colorectal that has spread to other parts of the body (metastatic). PolyPEPI1018 peptide vaccine is used to immunize against proteins present on the surface of tumor cells. This vaccine can activate the body's immune cells, called T cells. T cells fight infections and can also kill cancer cells. TAS-102 may help block the formation of growths that may become cancer. Giving PolyPEPI1018 and TAS-102 may kill more tumor cells in patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE I. To evaluate the safety and tolerability of multiple doses of colorectal cancer peptide vaccine PolyPEPI1018 (PolyPEPI1018) with trifluridine and tipiracil hydrochloride (TAS-102) in patients with metastatic colorectal cancer (mCRC).

SECONDARY OBJECTIVES:

I. To evaluate initial efficacy of PolyPEPI1018 with TAS-102 by evaluating progression free survival (PFS).

II. To evaluate initial efficacy of PolyPEPI1018 with TAS-102 by evaluating objective response rate (ORR).

III. To evaluate initial efficacy of PolyPEPI1018 with TAS-102 by evaluating duration of response (DoR).

IV. To evaluate initial efficacy of PolyPEPI1018 with TAS-102 by evaluating overall survival (OS).

CORRELATIVE OBJECTIVES:

I. Comparison of clinical benefit characteristics (ORR, PFS, OS or DoR) of the study with historical data of TAS-102.

II. Correlations between personal epitopes (PEPIs) identified by candidate CDx and T cell responses measured by enzyme-linked immune absorbent spot (ELISPOT).

III. To evaluate correlation between immune correlatives (T-cell responses in the blood and tumor and clinical benefit [ORR, PFS, OS or DoR]).

IV. To evaluate correlation between PEPIs/AGPs predicted by candidate CDx and clinical benefit (ORR, PFS, OS or DoR).

V. To evaluate the immunogenicity of PolyPEPI1018 by measuring both effector and memory T cell responses, VI. To evaluate immune activity of PolyPEPI1018 at tumor level (level of tumor infiltrating lymphocytes).

VII. To identify PEPIs (Personal EPItopes capable of inducing T cell responses in an individual) and AGPs (predicted number of expressed antigens likely hit by T cells) from PolyPEPI1018 in each patient.

OUTLINE:

Patients receive PolyPEPI1018 subcutaneously (SC) at 4 injection sites on days 1 and 15 and trifluridine and tipiracil hydrochloride orally (PO) twice daily (BID) on days 1-5 and 8-15. Treatment repeats every 28 days for up to 7 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Histologically confirmed metastatic adenocarcinoma originating from the colon or the rectum, microsatellite stable
* Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria

  * NOTE: Tumor lesions in a previously irradiated area are not considered measurable disease; Disease that is measurable by physical examination only is not eligible
* Received =< 2 lines of prior chemotherapy regimen for mCRC

  * NOTE: Adjuvant therapy will not be considered a line of therapy for mCRC unless the patient had disease recurrence =< 6 months of adjuvant therapy
* Provide written informed consent
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Absolute neutrophil count (ANC) >= 1500/mm^3 (obtained =< 21 days prior to registration)
* Platelet count >= 100,000/mm^3 (obtained =< 21 days prior to registration)
* Hemoglobin >= 9 g/dL (obtained =< 21 days prior to registration)
* Total bilirubin =< 1.5 x ULN (obtained =< 21 days prior to registration)
* Alanine aminotransferase (ALT) and aspartate transaminase (AST) =< 3 x ULN (=< 5 x ULN for patients with liver involvement) (obtained =< 21 days prior to registration)
* Calculated creatinine clearance >= 30 ml/min using the Cockcroft-Gault formula (obtained =< 21 days prior to registration)
* Anticipated life expectancy >= 6 months
* Negative urine pregnancy test done =< 7 days prior to registration, for persons of childbearing potential only

  * NOTE: If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Women of childbearing potential must agree to appropriately use an effective form of contraception (failure rate of < 1% per year) while enrolled in the study and for 3 months from the last vaccination. An effective form of contraception is defined as using hormonal contraceptives or an intrauterine device combined with at least 1 of the following forms of contraception: a diaphragm, cervical cap or condom
* Men must agree to use an effective form of contraception (as defined above), and not donate sperm for 3 months from the last vaccination
* Willingness to provide mandatory blood and buccal swab specimens for correlative research
* Willingness to provide mandatory tissue specimens for correlative research
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study). Note: During the active monitoring phase of a study

Exclusion Criteria:

* Received continuous systemic steroid treatment =< 2 weeks prior to registration
* Colorectal cancer with documented high microsatellite instability (MSI H)
* Pre-existing systemic autoimmune or antibody-mediated diseases or immune deficiency diseases
* Central nervous system (CNS) metastases
* Serious, non-healing wounds, ulcers or bone fractures
* Nephrotic syndrome
* Arterial thromboembolisms or severe hemorrhages =< 6 months before registration (except bleeding tumor before tumor resection surgery)
* Any of the following prior therapies:

  * Major surgery =< 12 weeks prior to registration or anticipation of needing such procedure during the study period
  * Radiation therapy =< 4 weeks prior to registration
  * Received chronic systemic immune therapy or immunosuppressant medication other than steroids =< 6 weeks prior to registration
* Uncontrolled pleural effusion, pericardial effusion or ascites requiring repeated drainage > once every 28 days
* Participants with active malignancy (other than colorectal cancer [CRC]) or a prior malignancy =< 12 months prior to registration

  * EXCEPTIONS: Non-melanotic skin cancer or carcinoma-in-situ of the cervix
* Acute or subacute intestinal obstruction or history of chronic intestinal inflammatory diseases
* Relevant toxicities of prior therapies must have resolved to =< grade 1, except for oxaliplatin-related neuropathy or alopecia
* Participant with myocardial infarction =< 6 months prior to registration or New York Heart Association Class III or IV, heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
* Administration of a live, attenuated vaccine =< 4 weeks prior to registration or anticipation of a live attenuated vaccine will be required during the study
* Participant has or will be participating in any of the following:

  * In another clinical study involving an investigational product (IP) or investigational device =< 30 days prior to registration or
  * Is scheduled to participate in another clinical study involving an IP or investigational device during the course of this study or
  * Is receiving any other investigational agent which would be considered as a treatment for colorectal cancer
* Known hypersensitivity to any component of the investigational drug
* Uncontrolled intercurrent non-cardiac illness including, but not limited to:

  * Ongoing or active infection
  * Psychiatric illness/social situations
  * Dyspnea at rest due to complications of advanced malignancy or other disease that requires continuous oxygen therapy
  * Any other conditions that would limit compliance with study requirements
* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant persons
  * Nursing persons
  * Men and women of childbearing potential who are unwilling to employ adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2023-06-11 (Actual); Study Completion 2023-06-11 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AE) | Up to 1 year
  The occurrence of at least 1 Grade 4 local AE or 1 Grade 3+ systemic AE during the first cycle of treatment. Evaluable patients are patients who are eligible, consented, received at least 50% of their expected cycle 1 trifluridine and tipiracil hydrochloride treatment, and received at least one dose of the PolyPEPI1018 Vaccine. The final local or systemic AE rate point estimate and corresponding 95% confidence interval will be reported.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 1 year
  ORR is defined as achieving complete response (CR) or partial response (PR) while on treatment. Disease status will be assessed using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria. ORR will be calculated as the proportion of evaluable patients who achieve response. The final ORR point estimate and corresponding 95% confidence interval will be reported.
Duration of response (DoR) | Up to 1 year
  DoR is defined at the time from first documented response (PR or CR) via RECIST 1.1 to progression or death. DoR will be estimated using the Kaplan-Meier method. Patients who are alive and progression-free will be censored at the last follow-up date. The median DoR and corresponding 95% confidence interval will be reported.
Overall survival (OS) | From registration to death from any cause, assessed up to 1 year
  OS will be estimated using the Kaplan-Meier method. Patients who are alive will be censored at the last follow-up date. The median OS and corresponding 95% confidence interval will be reported.
Progression free survival (PFS) | From registration to progression or death from any cause, whichever happens first, assessed up to 1 year
  Disease status will be assessed using RECIST 1.1 criteria. PFS will be estimated using the Kaplan-Meier method. Patients who are alive and progression-free will be censored at their last disease assessment date. The median PFS and corresponding 95% confidence interval will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Mojun Zhu, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

DOCUMENTS (1):
  • Informed Consent Form (2021-12-10): https://cdn.clinicaltrials.gov/large-docs/60/NCT05130060/ICF_000.pdf